CLINICAL TRIAL: NCT00576459
Title: A Randomized, Controlled Pilot Study to Evaluate the Safety and Efficacy of Intravitreal Fluocinolone Acetonide (0.5mg and 2mg) Implants in Patients With Clinically Significant Diabetic Macular Edema
Brief Title: Safety and Efficacy of Intravitreal Fluocinolone Acetonide Implants in Patients With Diabetic Macular Edema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 420-003
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-07

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Fluocinolone Acetonide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fluocinolone acetonide 0.59 mg (Experimental): 0.59 mg fluocinolone acetonide intravitreal implant
  Interventions: Drug: 0.59 mg fluocinolone acetonide intravitreal implant
- Fluocinolone acetonide 2.1 mg (Experimental): 2.1 mg fluocinolone acetonide intravitreal implant
  Interventions: Drug: 2.1 mg fluocinolone acetonide intravitreal implant
- Laser photocoagulation (Active Comparator): standard of care laser photocoagulation
  Interventions: Procedure: standard of care laser photocoagulation

INTERVENTIONS:
Drug: 0.59 mg fluocinolone acetonide intravitreal implant — 0.59 mg
  Other Names: Retisert
  Arms: Fluocinolone acetonide 0.59 mg
Drug: 2.1 mg fluocinolone acetonide intravitreal implant — 2.1 mg
  Arms: Fluocinolone acetonide 2.1 mg
Procedure: standard of care laser photocoagulation — standard of care laser photocoagulation
  Arms: Laser photocoagulation

SUMMARY:
This is a 3-year randomized, dose masked, three-arm controlled, pilot study to evaluate the safety and efficacy of the intravitreal FA implants (0.59mg and 2.1mg), when compared to laser photocoagulation in the treatment of patients with diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 1 or 2 diabetes.
* Subjects with clinically significant macular edema as defined by the ETDRS.
* A best corrected visual acuity between +0.30 and +1.00 logMAR (70 and 35 letters or approximately 20/40 to 20/200) as measured on an ETDRS chart.
* Subjects with laser treatment status/history as follows: [1] Naïve to laser photocoagulation or Focal laser photocoagulation more than 16 weeks prior to screening or PRP more than 24 weeks prior to screening, [2] No laser scars within 500µm (4x the width of a retinal vein at the disc margin) of the central macula.
* The subject's ocular media had to be sufficiently clear to allow for quality fundus photography.
* If aphakic or pseudophakic, lens removal had to have occurred at least 40 weeks prior to screening.
* Subjects had to be males or non-pregnant females of at least 18 years.
* Subjects had to display the ability and willingness to comply with treatment, follow up process, and sign an Informed Consent Form.

Exclusion Criteria:

* Subjects who have had previous grid macular photocoagulation for diffuse macular edema.
* Presence of posterior hyaloid membrane, epiretinal membranes, fibrovascular proliferation, and vitreopapillary traction, which causes tractional distortion on the macula as demonstrated by OCT or funduscopy.
* History of or current retinal detachment requiring surgical treatment or a scleral buckle.
* Diabetic Retinopathy that required immediate PRP.
* Ocular disease other than diabetic retinopathy that could confound the outcome of the study (e.g., age-related macular degeneration, drug toxicity, uveitis, hypertensive retinopathy, ischemic maculopathy, etc.).
* Glaucoma, or history of glaucoma in either the study eye or the fellow eye.
* Ocular hypertension, or history of ocular hypertension requiring IOP lowering treatment.
* A media opacity that precludes visualization and/or diagnosis of the status of the eye.
* Concurrent coumadin therapy or known bleeding diathesis.
* Subjects requiring chronic systemic corticosteroid therapy or systemic immunosuppressive therapy to manage non-ocular disease.
* Concurrent treatment with a new investigational drug.
* Subjects with a best-corrected visual acuity worse than +1.0 logMAR (20/200 or 35 ETDRS letters) in the fellow eye.
* Pregnant or lactating females.
* Females of childbearing potential considering becoming pregnant during the course of the study and those not taking effective contraception/precautions to avoid pregnancy.
* History of hypersensitivity to fluorescein, known allergies to steroids or any component of the intraocular device.
* Subjects with photophobia that will preclude the ability to do fundus evaluations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2003-03; Primary Completion 2006-06 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Between group difference in mean visual acuity change (from baseline) | 1 year

SECONDARY OUTCOMES:
Differences in the proportions of subjects in each treatment group experiencing changes in: the area of retinal thickening; retinal leakage and cystoid scores; grade of diabetic retinopathy | 1 year
Ocular adverse events, non-ocular adverse events, and intraocular pressure >/= 30 mm Hg | throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Taraprasad Das, MD, Principal Investigator — LV Prasad Eye Institute; Dennis Lam Shun-Chiu, MD, Principal Investigator — Chinese University of Hong Kong
Locations (2):
- The Chinese University of Hong Kong, Hong Kong, China
- LV Prasad Eye Institute, Banjara Hills, Hyderabad, India